CLINICAL TRIAL: NCT05883735
Title: Retrospective Study of Radio-induced Toxicities in the Treatment of Lung Cancer With Tomotherapy
Acronym: ETRICAPT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-05Obs-CHRMT
Record Dates: First submitted 2023-05-19; First posted 2023-06-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Tomotherapy; Toxicity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancers treated by Tomotherapy represent between 60 and 100 patients per year at the CHR of Metz-Thionville. Some patients were observed to present acute toxicities during treatment such as dysphagia or esophagitis of CTCAE grade > 2. Beyond well known therapeutic and comorbidities factors, the pathophysiology of these events is largely ruled by a constitutional factor - the enzymatic equipment allowing more or less good repair of the DNA lesions induced by radiotherapy (RT). This equipment is characteristic of each individual, hence the term individual radiosensitivity (IR).The scientific literature is rather poor in data describing the frequency of these toxicities in patients receiving RT for lung cancer.

The objective of this study is to describe the frequency of acute and late toxicities after normofractionated radiotherapy of 66 Gy in 33 fractions in patients with small cell or non-small cell lung cancer, stage 2 or 3.

ELIGIBILITY:
Inclusion Criteria:

* stage II-III non-small cell or small cell lung cancer treated with normo-fractionated radiotherapy of 66Gy in 33 fractions using Tomotherapy

Exclusion Criteria:

* patient who refused to be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will consist of patients with stage II-III non-small cell or small cell lung cancer (ICD-10 code: C34) treated with normo-fractionated radiotherapy of 66 Gy in 33 fractions using Tomotherapy between January 2016 and April 2023 at CHR Metz-Thionville.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
late toxicity of radiotherapy | up to 2 years after tomotherapy treatment
  according to CTCAE v5.0 grading

SECONDARY OUTCOMES:
acute toxicity of radiotherapy | 6 months following tomotherapy treatment
  according to CTCAE v5.0 grading

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MICHEL, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France